CLINICAL TRIAL: NCT06992154
Title: Acne Treatment With Akkermansia Muciniphila, Clostridium Beijerinckii, Anaerobutyricum Hallii, Clostridium Butyricum, Bifidobacterium Infantis Probiotic Capsule to Impact Metabolic Health
Brief Title: Role of Akkermansia Muciniphila in Acne Vulgaris
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00137381
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Probiotic Group (Experimental): Participants will receive a 12-week probiotic course.
  Interventions: Dietary Supplement: Akkermansia Muciniphila, Clostridium Beijerinckii, Anaerobutyricum Hallii, Clostridium Butyricum, Bifidobacterium Infantis Probiotic Capsule

INTERVENTIONS:
Dietary Supplement: Akkermansia Muciniphila, Clostridium Beijerinckii, Anaerobutyricum Hallii, Clostridium Butyricum, Bifidobacterium Infantis Probiotic Capsule — Probiotic capsule will contain Akkermansia Muciniphila, Clostridium Beijerinckii, Anaerobutyricum Hallii, Clostridium Butyricum, and Bifidobacterium Infantis

SUMMARY:
The project explores the use of Pendulum's Glucose Control, which contains a unique combination of probiotics, including Akkermansia muciniphila, Clostridium beijerinckii, Anaerobutyricum hallii, Clostridium butyricum, and Bifidobacterium infantis, to treat acne by improving gut health and reducing inflammation. These probiotic strains work synergistically to enhance the gut's protective barrier, lower harmful substances such as lipopolysaccharides, and increase the production of beneficial compounds like short-chain fatty acids, which can help modulate immune response and inflammation associated with acne. By integrating this probiotic combination into treatment strategies, the approach aims to offer a natural and effective solution for clearer skin. Additionally, the project seeks to investigate the correlation between postprandial glucose spikes and acne flare-ups. Continuous glucose monitoring (CGM) will be employed to track blood glucose fluctuations following meals, providing valuable insights into the potential link between metabolic responses and acne severity. This comprehensive approach aims to enhance understanding of how gut health, inflammation, and metabolic factors interact in the context of acne management.

DETAILED DESCRIPTION:
Akkermansia muciniphila, Clostridium beijerinckii, Anaerobutyricum hallii, Clostridium butyricum, and Bifidobacterium infantis are emerging as promising candidates for next-generation probiotics with potential applications in the management of acne. These microorganisms have been recognized for their roles in enhancing gut barrier function and contributing to a healthy gut microbiota composition. Through mechanisms such as strengthening the gut mucosal barrier and reducing systemic lipopolysaccharide levels, these probiotics may help mitigate systemic inflammation and lower inflammatory markers. Additionally, their capacity to produce short-chain fatty acids, including acetate, propionate, and butyrate, may contribute to immune modulation and a reduction in inflammatory processes, which are relevant to acne pathogenesis. This evidence highlights the potential utility of these probiotics in therapeutic strategies aimed at improving acne outcomes via modulation of the gut microbiota.

In this study, investigators also aim to explore the relationship between postprandial glucose spikes and acne flare-ups. To investigate this, investigators will utilize continuous glucose monitoring (CGM) to track fluctuations in blood glucose levels following meals. By correlating these glucose spikes with changes in acne severity, investigators hope to gain a deeper understanding of the potential connection between metabolic responses and inflammatory skin conditions. This approach will provide valuable insight into how dietary factors and gut microbiota modulation may interact to influence acne outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 45 years.
* Individuals with clinically diagnosed moderate to severe acne vulgaris, determined using standardized scales like the Global Acne Grading
* System (GAGS) by Investigators of the study.
* Willingness to provide informed consent and adhere to study protocols, including follow-ups and sample collections.

Exclusion Criteria:

* Recent and/or current antibiotic use: Individuals who have used antibiotics or probiotics within the last three months, as these can alter gut microbiota composition
* Chronic gastrointestinal conditions: Participants with chronic gastrointestinal conditions such as Chron's disease, ulcerative colitis or irritable bowel syndrome (IBS).
* Immune disorders: Individuals with known immune deficiencies or autoimmune diseases, which might affect inflammation levels and study outcomes.
* Pregnancy or Lactation: pregnant or breastfeeding women, due to potential risk and hormonal changes that could influence acne and gut health.
* Inability or unwillingness of subject or legal guardian/representative to give informed consent
* Oral acne medications, including isotretinoin and spironolactone: these medications can significantly alter acne severity, making it difficult to isolate and accurately measure the effects of the probiotic intervention. Isotretinoin, a powerful retinoid, and spironolactone, a hormone-modulating medication, both have well-documented impacts on acne that could confound the study's results. Excluding participants using these medications ensures that changes in acne severity can be more directly attributed to the probiotic being tested, leading to clearer, more reliable findings on its efficacy.
* History of metabolic disorders such as type 1 diabetes (DM1) and type 2 diabetes (DM2): DM1 and DM2 and their therapies can significantly alter baseline metabolic markers, such as glucose levels, insulin sensitivity, and inflammatory responses. Including such individuals might confound the results and make it difficult to attribute observed effects solely to the probiotics.
* Chronic gastrointestinal conditions: Participants with chronic gastrointestinal conditions such as Crohn's disease, ulcerative colitis or irritable bowel syndrome (IBS).
* Known hypersensitivity to >4 first-line antimicrobial therapies against Akkermansia muciniphila, Clostridium beijerinckii, Clostridium butyricum, Anaerobutyricum hallii: Penicillin, Piperacillin, Tetracycline, Amoxicillin, Ampicillin
* Known hypersensitivity to >4 first-line antimicrobial therapies against Bifidobacterium infantis Bi-26TM: Gentamicin, Kanamycin, Streptomycin, Tetracycline, Erythromycin, Clindamycin, Ampicillin, Vancomycin
* Known allergy or hypersensitivity to any of the following ingredients: Akkermansia muciniphila, Anaerobutyricum hallii, Bifidobacterium infantis, Clostridium beijerinckii, and Clostridium butyricum Other Ingredients: Chicory inulin and oligofructose (prebiotic fiber), hypromellose (vegetarian capsule), fruit & vegetable juice (coloring agent), magnesium stearate (flow agent for encapsulation), and silica.
* Immune disorders: Individuals with known immune deficiencies or autoimmune diseases, which might affect inflammation levels and study outcomes.
* BMI of greater than or equal to 45: Excess adiposity is likely to impact sex hormones, inflammation, insulin resistance, and GLP-1 levels. These factors could confound the study outcomes. Additionally, excess adiposity is associated with hyperandrogenism and changes in sex hormone-binding globulin (SHBG), which may independently influence acne severity and skew results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acne severity reduction | 12 weeks
  The primary outcome measure will be the reduction in acne severity from baseline, as assessed by a validated acne severity scoring system (the Global Acne Grading System). Acne severity will be evaluated based on the number, type, and distribution of lesions, as well as the overall clinical assessment of the skin condition. Assessments will be conducted at baseline and specified follow-up intervals to determine the extent of improvement. Reduction in severity will be quantified as a percentage change from baseline scores.

SECONDARY OUTCOMES:
Association Between Postprandial Glucose Spikes and Acne Flares | 12 weeks
  The secondary outcome measure will evaluate the association between postprandial glucose spikes and the frequency or severity of acne flares. Postprandial glucose levels will be monitored using continuous glucose monitoring at designated intervals. Acne flares will be assessed using a validated acne severity scoring system along with participant journals, with flare frequency and changes in lesion count/type recorded over the study period. Correlations between glucose spike magnitude and acne flare characteristics will be analyzed to identify potential relationships.